CLINICAL TRIAL: NCT06586762
Title: Symmetry in Sagittal Knee Kinematics of Transtibial Amputee: Daily-Use Prosthesis Vs Running-Specific Prosthesis
Brief Title: Sagittal Knee Kinematics of Transtibial Amputee with Running Blade
Status: Completed | Type: Observational
Sponsor: Baskent University (Other)
Collaborators: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, Senay Cerezci Duygu, Asst. Prof., Istanbul Saglik Bilimleri University
Other Study IDs: 2024/369
Record Dates: First submitted 2024-09-02; First posted 2024-09-19 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2024-09

CONDITIONS: Amputation; Prosthesis User
Keywords: amputee; symmetry; knee; running; running-specific prosthesis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Daily-Use Prosthesis (DUP): Participants are going video recorded in the sagittal plane, to convert knee flexion motion into angles for the amputated and intact knee and to make measurements using the software's virtual goniometer. The recording will be taken during walking at self-selected walking speed with DUP.
- Running-Specific Prosthesis (RSP): Participants are going video recorded in the sagittal plane, to convert knee flexion motion into angles for the amputated and intact knee and to make measurements using the software's virtual goniometer. The recording will be taken during slow-running (heel-strike jogging) with RSP.

SUMMARY:
Introduction: People with transtibial amputation often suffer musculoskeletal deformities in the form of knee osteoarthritis or osteophytosis due to asymmetric movement patterns and often complain of associated symptoms. Therefore, this study aims to evaluate the sagittal kinematics of the intact and residual knee in the use of Running-Specific Prostheses (RSP), which are increasing in popularity and use among amputees.

Materials and Methods: Participants will be video recorded in the sagittal plane to convert knee flexion motion into angles for the amputee and intact knee and to make measurements using the software's virtual goniometer. Recordings will be taken under the following two conditions: 1) walking at a self-selected walking speed with a Daily Use Prosthesis (DUP); 2) Slow running with RSP. The peak flexion during the swing phase and the initial flexion during the first contact of the stance phase will be recorded as angles in both conditions.

ELIGIBILITY:
Inclusion Criteria:

* body mass index below 30 kg/m2,
* Having unilateral transtibial amputation,
* Being at K4 functional level,
* Having an existing running blade,
* Being able to use RSP integrating it into their DUP,
* Having no self-reported problems with the residual limb or prosthesis, pain or skin lesions,
* Being active recreational runners (at least once a week) for at least 1 and up to 3 months without injury.

Exclusion Criteria:

* Having a history of knee surgery or contracture in the intact/amputee knee.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Unilateral transtibial amputee at K4 functional level
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2024-09-05 (Actual); Primary Completion 2024-10-05 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Sagital Knee Kinematics of intact and residual knee with Daily-Use Prosthesis (DUP) | Baseline
  In the sagittal plan, knee flexion motion for the amputated and intact knee will be recorded during walking at self-selected walking speed with Daily-Use Prosthesis (DUP). The peak flexion during swing phase and the initial flexion during initial contact of the stance phase were recorded as angle.
Sagital Knee Kinematics of intact and residual knee with Running-Specific Prosthesis (RSP) | Same day as baseline; 10 minutes after RSP integrated to prosthesis.
  In the sagittal plan, knee flexion motion for the amputated and intact knee will be recorded during slow-running (jogging) with Running-Specific Prosthesis (RSP). The peak flexion during swing phase and the initial flexion during initial contact of the stance phase were recorded as angle.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Ankara, Etlik Keçiören, Turkey (Türkiye)